CLINICAL TRIAL: NCT00763373
Title: Unnecessary IV Antibiotic Days Using General Criteria for Antibiotic Switch
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Bjoern Waagsboe, Sorlandet Sykehus HF
Other Study IDs: Antibiotic Switch
Record Dates: First submitted 2007-08-16; First posted 2008-09-30 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Infection
Keywords: Lower respiratory infection; Upper respiratory infection; Urinary tract infection; Soft tissue infection; Hepatobiliary infection
MeSH Terms: conditions — Infections; Respiratory Tract Infections; Urinary Tract Infections; Soft Tissue Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Observation group
- 2: Intervention group
  Interventions: Other: Implementation of antibiotic switch guidelines

INTERVENTIONS:
Other: Implementation of antibiotic switch guidelines — Implementation of antibiotic switch guidelines
  Other Names: Antibiotic switch
  Groups: 2

SUMMARY:
Observation of the use of intravenous antibiotics in medical clinic of Sorlandet Hospital, Norway. Suggestions of criteria for the switch from intravenous to oral administration of antibiotics. Implementation of the criteria and new registration of the use of intravenous antibiotics. Comparison of the amount of the iv-administration before and after the intervention.

DETAILED DESCRIPTION:
The study is a comparison of the use of intravenous antibiotics before and after the implementation of switch criteria. Switch is defined as a change in administration route from intravenous to oral.

Patients administered to medical department at Sorlandet hospital in Kristiansand and Arendal are included if they are receiving intravenous antibiotics. Pediatric department is not included. Patients that are already hospitalized and given intravenous antibiotics are also included.

Patients that are excluded are those with CNS-infection, endocarditis, bone/joint infection, deep undrainable abscesses and those with foreign body infection.

Switch criteria are made from a thorough investigation on earlier switch studies. We have collected several studies on this topic, but none from the nordic countries.

The intervention contributes the following: The implementation of a registration form where doctors are prone to answer six questions when they evaluate antibiotic administration form.

1. Are there special iv-indications? (CNS-infection, endocarditis, bone/joint infection, deep undrainable abscesses or foreign body infection)
2. Is the oral route compromized? (unconscious, nausea, vomiting, diarrhoea, dysphagia, lack of cooperativeness)
3. Is the patients suffering from immunosuppression? (leukopenia, cytotoxic treatment, transplantation, steroids >10mg, TNF-alfa inhibitor treatment, unregulated diabetes mellitus (HbA1C >10), uremia (serum-creatinine > 300), HIV, AIDS, lymphoma, multiple myelomas, cystic fibrosis, asplenic)
4. Is the systemic inflammatory response syndrome present?
5. Is the preferred antibiotics only available in intravenous form?
6. Are there any other special reasons for intravenous antibiotics?

If the doctor can answer NO to all these questions, then the patient is a candidate for antibiotic switch from day three after hospitalization. This evaluation form follows the other medical registration forms from day to day.

The intervention also includes

* A lecture by the study group to all our medical doctors.
* Information by e-mail to all our medical doctors
* Information by letters to all our medical doctors and chief nurses

Registration of parameters used for evaluating antibiotic switch is done three times a week by the study group. We register date and patient information, if other medication is taken orally, heart rate, respiratory rate, temperature, biochemical parameters (CRP and leukocytes), diagnosis and antibiotic choice.

ELIGIBILITY:
Inclusion Criteria:

* Alle patients with suspected infection and who is gives intravenous antibiotics

Exclusion Criteria:

* CNS-infection
* Endocarditis
* Bone/joint infection
* Undrained abscess
* Foreign body infection
* Compromized oral route
* Immunosuppression
* Patients meeting the systemic inflammatory response syndrome criteria
* No preferred oral antibiotic available
* Other conditions requiring intravenous administration

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2006-11; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Reduction in the amount of intravenous antibiotic days | During stay

SECONDARY OUTCOMES:
Hospital stay duration, re-admittance, re-prescription of intravenous antibiotic therapy | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bjoern Waagsboe, Ass dr, Principal Investigator — Medical department Kristiansand; Anders Sundoy, Chief Doc, Study Director — Medical dep kristiansand; Else Quist Paulsen, ass doc, Study Director — Med dep Arendal
Locations (2):
- Norway (2):
  - Sorlandet Sykehus Arendal, Arendal, Aust-Agder
  - Sørlandet Sykehus Kristiansand, Kristiansand, Vest Agder